CLINICAL TRIAL: NCT03709173
Title: FuRST 2.0: Cognitive Pre-testing for a New Functional Rating Scale for Use in Huntington's Disease - Round 2
Brief Title: FuRST 2.0 Cognitive Pre-testing - Round 2
Status: Completed | Type: Observational
Sponsor: CHDI Foundation, Inc. (Other)
Collaborators: Dr. Glenn T. Stebbins (Rush University Medical Center ) (Unknown); Dr. Nancy LaPelle (Unknown)
Responsible Party: Sponsor
Other Study IDs: C-000918-3
Record Dates: First submitted 2018-09-25; First posted 2018-10-17 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Premanifest HDGEC participants
  Interventions: Behavioral: FuRST 2.0
- Early-manifest HDGEC participants
  Interventions: Behavioral: FuRST 2.0
- Companions of Premanifest HDGEC
  Interventions: Behavioral: FuRST 2.0
- Companions of Early-manifest
  Interventions: Behavioral: FuRST 2.0

INTERVENTIONS:
Behavioral: FuRST 2.0 — Round 2 of cognitive pre-testing for a new functional rating scale

SUMMARY:
The study is a single, cross-sectional cognitive interview of FuRST 2.0, functional rating scale, administered to forty Huntington's Disease Gene Expansion Carriers (HDGECs) and potentially, their companions (the companion's participation is optional in this study). The scale will be tested as a patient reported outcome (PRO) in that the information will come directly from the HDGEC participant or the HDGEC participant together with his/her companion through self-report. The purpose is to identify real or potential comprehension or usage problems with scale items, response options, instructions and disclaimer statement, which are all components of the FuRST 2.0 scale. Through a structured cognitive interview with the HDGEC participants or the HDGEC participants together with their companions, followed by qualitative analysis, the final phrasing of the individual scale items, response options, instructions and disclaimer statement for the scale will be generated. Depending on the results of this study, an additional round of cognitive pre-testing may be required in a separate study.

ELIGIBILITY:
Inclusion Criteria for Premanifest HDGECs:

* Identified as an active participant in Enroll-HD (participants who have completed their last onsite Enroll-HD visit within approximately 15 months)
* At least 18 years of age
* Fluent in English and had his/her primary education in English
* Able and willing to provide critical feedback (per site PI or site PI's designee discretion)
* Willing and able to provide written informed consent
* Cytosine, Adenine, Guanine (CAG) length ≥ 40
* Disease burden score (DBS) ≥ 250
* Diagnostic confidence level (DCL) ≤ 3

Inclusion Criteria for Early-manifest HDGECs:

* Identified as an active participant in Enroll-HD (participants who have completed their last onsite Enroll-HD visit within approximately 15 months)
* At least 18 years of age
* Fluent in English and had his/her primary education in English
* Able and willing to provide critical feedback (per site PI or site PI's designee discretion)
* Willing and able to provide written informed consent
* CAG length ≥ 36
* DCL= 4
* Total Functional Capacity (TFC) ≥11

Inclusion Criteria for a Companion of an HDGEC

* At least 18 years of age
* Fluent in English and had his/her primary education in English
* In his/her opinion, has sufficient interaction and knowledge of the HDGEC participant's capabilities and daily activities
* Is acceptable to the HDGEC participant and the site PI or site PI's designee
* Willing and able to provide written informed consent

Exclusion Criteria for an HDGEC/a companion of HDGEC:

* Significant cognitive or any other impairment sufficient to interfere with study associated tasks as judged by the site PI or the site PI's designee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An HDGEC: Premanifest and early-manifest HDGEC who is also a participant in Enroll-HD and meets the protocol selection criteria for the HDGEC. HDGEC participants will be recruited from English speaking Enroll-HD sites.
  A Companion: A person who, in his/her opinion, has sufficient interaction and knowledge of the HDGEC participant's capabilities and daily activities, is acceptable to the HDGEC participant and the site principal investigator (site PI) or site PI's designee and meets the protocol selection criteria for the companion. The companion's participation is optional in this study.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2019-08-02 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Participant's comprehension of the FuRST 2.0 rating scale measured by qualitative analysis. | 7 months
  The primary assessment will use qualitative analysis of the cognitive interview to determine the usability of the FuRST 2.0 scale in the HD population.
  Note: The instructions, items, response options and disclaimer statement are all part of the FuRST 2.0 scale.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Rocky Mountain Movement Disorders Center, P.C., Englewood, Colorado
  - Hereditary Neurological Disease Centre, Inc., Wichita, Kansas
  - Columbia University, New York, New York
- Centre for Movement Disorders (Neuropharm Consulting), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided